CLINICAL TRIAL: NCT06271967
Title: A Study of FOCAL Pulsed Field Ablation With the TactiFLEX SE Catheter and Volt Generator for the Treatment of Paroxysmal Atrial Fibrillation (FOCALFLEX)
Brief Title: FOCALFLEX (CE Mark) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10518
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation Paroxysmal
Keywords: Pulse Field Ablation; Ablation Catheter; arrhythmia; PFA; Paroxysmal AF
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- treatment arm (Experimental): Patients treated for paroxysmal atrial fibrillation with the TactiFlex™ Ablation Catheter Sensor Enabled™ (SE).
  Interventions: Device: TactiFlex™ Ablation Catheter Sensor Enabled™

INTERVENTIONS:
Device: TactiFlex™ Ablation Catheter Sensor Enabled™ — Pulsed field ablation (PFA)/radiofrequency (RF) ablation with the TactiFlex™ Ablation Catheter Sensor Enabled™

SUMMARY:
This clinical investigation is intended to demonstrate safety and effectiveness of the TactiFlex™ Ablation Catheter Sensor Enabled™, the Volt™ Pulse Field Ablation (PFA) Generator, and EnSite™ X EP System with EnSite™ Pulsed Field Ablation Software for the treatment of symptomatic, recurrent paroxysmal atrial fibrillation (PAF).

DETAILED DESCRIPTION:
This is a pre-market, prospective, single-arm, non-randomized, multicenter clinical investigation. Up to 150 subjects will be enrolled in this clinical investigation at up to 25 investigational sites worldwide. The clinical investigation is sponsored by Abbott.

ELIGIBILITY:
Inclusion Criteria:

1. Documented symptomatic paroxysmal AF (PAF). Documentation requirements are as follows:

   1. Physician's note indicating recurrent self-terminating AF with ≥ 2 episodes of PAF within the 6 months prior to enrollment AND
   2. One electrocardiographically documented PAF episode within 12 months prior to enrollment.
2. Plans to undergo a catheter ablation procedure due to symptomatic PAF
3. At least 18 years of age
4. Able and willing to comply with all trial requirements including pre-procedure, post- procedure, and follow-up testing and requirements
5. Informed of the nature of the trial, agreed to its provisions, and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee (IRB/EC) of the respective clinical trial site.

Exclusion Criteria:

1. Previously diagnosed persistent or long-standing persistent atrial fibrillation (Continuous AF greater than 1 year in duration)
2. Arrhythmia due to reversible causes including thyroid disorders, acute alcohol intoxication, electrolyte imbalance, severe untreated sleep apnea, and other major surgical procedures in the preceding 90 days
3. Known presence of cardiac thrombus
4. Left atrial diameter (LAD) ≥ 5.5 cm (anteroposterior diameter) within 180 days prior to the index procedure
5. Left ventricular ejection fraction (LVEF) < 35% as assessed with echocardiography or computerized tomography (CT) within 180 days prior to the index procedure
6. New York Heart Association (NYHA) class III or IV heart failure
7. Body mass index > 40 kg/m2
8. Pregnant or nursing
9. Patients who have had a ventriculotomy or atriotomy within the preceding 28 days of procedure
10. Myocardial infarction (MI), acute coronary syndrome, percutaneous coronary intervention (PCI), or valve or coronary bypass grafting surgery within preceding 90 days
11. Stroke or TIA (transient ischemic attack) within the last 90 days
12. Heart disease in which corrective surgery is anticipated within 180 days after procedure
13. History of blood clotting or bleeding abnormalities including thrombocytosis, thrombocytopenia, bleeding diathesis, or suspected anti-coagulant state
14. Contraindication to long term anti-thromboembolic therapy
15. Patient unable to receive heparin or an acceptable alternative to achieve adequate anticoagulation
16. Known sensitivity to contrast media (if needed during the procedure) that cannot be controlled with pre-medication
17. Previous left atrial surgical or left atrial catheter ablation procedure (including left atrial appendage (LAA) closure device)
18. Plans to have an LAA closure device implanted during the follow-up period
19. Presence of any condition that precludes appropriate vascular access
20. Severe mitral regurgitation (regurgitant volume ≥ 60 mL/beat, regurgitant fraction ≥ 50%, and/or effective regurgitant orifice area ≥ 0.40cm2).
21. Previous tricuspid or mitral valve replacement or repair
22. Patients with prosthetic valves
23. Patients with a myxoma
24. Patients with an interatrial baffle or patch as the transseptal puncture could persist and produce an iatrogenic atrial shunt
25. Stent, constriction, or stenosis in a pulmonary vein
26. Rheumatic heart disease
27. Hypertrophic cardiomyopathy
28. Active systemic infection
29. Renal failure requiring dialysis
30. Severe pulmonary disease (e.g., restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces severe chronic symptoms
31. Presence of an implantable therapeutic cardiac device including permanent pacemaker, biventricular pacemaker, or any type of implantable cardiac defibrillator (with or without biventricular pacing function) or planned implant of such a device for any time during the follow-up period. Presence of an implantable loop recorder is acceptable as long as it is removed prior to insertion of the investigational device.
32. Patient is currently participating in another clinical trial or has participated in a clinical trial within 30 days prior to screening that may interfere with this clinical trial without pre-approval from this study Sponsor
33. Unlikely to survive the protocol follow up period of 12 months
34. Presence of other medical, anatomic, comorbid, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
35. Individuals without legal authority
36. Individuals unable to read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2026-01-19 (Actual)

PRIMARY OUTCOMES:
Incidence of primary safety endpoint events | 7 days
  The primary safety endpoint is the proportion of subjects experiencing a device and/or procedure-related serious adverse event (SAE) with onset within 7 days of any ablation procedure (index or repeat procedure performed 0-90 days post initial procedure) that uses the TactiFlex PFA System defined below:
  * Atrio-esophageal fistula
  * Cardiac tamponade/perforation
  * Death
  * Heart block
  * Myocardial infarction
  * Pericarditis
  * Phrenic nerve injury resulting in diaphragmatic paralysis
  * Pulmonary edema
  * Pulmonary vein stenosis
  * Stroke/cerebrovascular accident
  * Thromboembolism
  * Transient ischemic attack
  * Vagal nerve injury/gastroparesis
  * Major Vascular access complications / major bleeding event
  * Device and/or procedure related cardiovascular and/or pulmonary adverse event that prolongs hospitalization for more than 48 hours (excluding hospitalization solely for arrhythmia recurrence or non-urgent cardioversion)
Freedom from documented AF/AFL/AT recurrence | 6 months
  The primary effectiveness endpoint for this clinical trial is freedom from documented (symptomatic or asymptomatic) AF/AFL/AT episodes of >30 seconds duration that are documented by protocol-specified 12-lead ECG, TTM or Holter monitor (HM) devices after the index ablation procedure through 6 months of follow-up (after a 90-day blanking period following the index ablation procedure).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kammer, Study Director — Abbott
Locations (24):
- Australia (4):
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, Saustrl
  - Peninsula Private Hospital, Langwarrin, Victoria
  - Royal Melbourne Hospital - City Campus, Parkville, Victoria
- Austria (2):
  - Universitätsklinik Graz, Graz, Styria
  - A. ö. Krankenhaus der Elisabethinen Linz, Linz, UPR AUS
- UZ Brussel, Brussels, B CAP R, Belgium
- Nemocnice Ceske Budejovice, a.s., České Budějovice, Sbohmia, Czechia
- Skejby University Hospital, Aarhus, Arhus, Denmark
- France (3):
  - Hopital Haut Leveque, Pessac, Aquitaine
  - CHU Trousseau, Chambray-lès-Tours, Centre-Val de Loire
  - Hôpital Pitié Salpetrière, Paris, ILE
- Germany (2):
  - Deutsches Herzzentrum München des Freistaates Bayern, München, Bavaria
  - Herz-und Diabetes Zentrum NRW, Bad Oeynhausen, N. RHIN
- Italy (2):
  - Ospedale San Raffaele, Milan, Lombard
  - Centro Cardiologico Monzino, Milan, Lombard
- Netherlands (4):
  - Universitair Medische Centrum Groningen, Groningen, Grogen
  - St. Antonius Ziekenhuis, Nieuwegein, Utrecht
  - Leiden University Medical Center, Leiden, Zuid
  - Haga Ziekenhuis Locatie Leyenburg, The Hague, ZUID
- Spain (3):
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari i Politècnic La Fe, Valencia, Valncia
- The Royal Sussex County Hospital, Brighton, Soeast, United Kingdom

IPD SHARING:
Plan to Share IPD: No